CLINICAL TRIAL: NCT03624049
Title: The Impact of Expanding a Community-Based Exercise Program on Social Connectedness and Falls Prevention in Older Adults: Leveraging Exercise to Age in Place (LEAP)
Brief Title: The Impact of Community Exercise on Social Connectedness and Falls in Older Adults: Leveraging Exercise to Age in Place
Acronym: LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Jewish Family Service (Unknown); Partners In Care Foundation (Unknown); AARP Foundation (Other)
Responsible Party: Principal Investigator, Allison Mays, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro51676
Record Dates: First submitted 2018-07-12; First posted 2018-08-09 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Social Isolation; Fall
MeSH Terms: conditions — Social Isolation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pre-post study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Exercise Program (Other): Participation in Health Class including: Arthritis Exercise Foundation Exercise Class, Tai Chi for Arthritis, EnhanceFitness Class, or Healthier Living Class.
  Interventions: Other: Exercise; Other: Health Class

INTERVENTIONS:
Other: Exercise — Community based exercise programs held 2-3 times per week
Other: Health Class — Community based health class held 1 time per week

SUMMARY:
The goal of this study is to reduce risk of falls and social isolation in older adults age 50+ through participation in community based health and exercise programs.

DETAILED DESCRIPTION:
PRIMARY HYPOTHESES: In community-dwelling ambulatory older adults (age ≥50 years) participation in a community-based group program will improve the Duke Social Support Index (DSSI) score by four points measured after six to eight participation in the program when compared to the DSSI score prior to participation in the program. This increase will be sustained at 26 week follow-up.

SECONDARY HYPOTHESES: Participants in the community-based group exercise activities will have decreased fall risk when measured after six to eight weeks participation in the program when compared to pre-participation as based on responses to the fall risk questionnaire. Cedars-Sinai patients who participate in the community-based programs will have a decrease in health care utilization (as measured by physician visits, Emergency Department visits, and hospitalizations) in the 26 weeks after program enrollment compared to the 26 weeks prior to program enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Must be cognitively stable and must be 50 years or older

Exclusion Criteria:

* <50 years
* Cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Social Isolation | Change in Duke Social Support Index from baseline will be measured at 8 weeks and 6 months.
  The Duke Social Support Index (DSSI) is an 11 item questionnaire with a total score between 11 and 33 with higher scores indicating increased social connection and lower scores indicating higher social isolation.

SECONDARY OUTCOMES:
Number of falls in the past 3 months - Reduce Falls | Items will be measured at Baseline, 8 weeks, and 6 months
  Number of falls in the past 3 months
Number of falls with injury in the past 3 months - Reduce Falls | Items will be measured at Baseline, 8 weeks, and 6 months
  Number of falls with injury in the past 3 months
Change in Loneliness | Items will be measured at Baseline, 8 weeks, and 6 months; assessing a change in loneliness from baseline to 8 weeks and 6 months
  University of California Los Angeles 3 item Loneliness scale is a 3 item questionnaire with a total score between 3 and 9 with higher scores indicating increased loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Mays, MD, Principal Investigator — Cedars-Sinai Medical Center; Sonja Rosen, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (9):
- United States (9):
  - Roxbury Park Community Center, Beverly Hills, California
  - Washington Irving Branch Library, Los Angeles, California
  - Pan Pacific Park, Los Angeles, California
  - People Coordinated Services- Crenshaw, Los Angeles, California
  - Poinsettia Park, Los Angeles, California
  - Will and Ariel Durant Library, Los Angeles, California
  - Virtual recruiting, Los Angeles, California
  - Yvonne B. Burke Senior & Community Center, Los Angeles, California
  - West Hollywood Park Auditorium, West Hollywood, California